CLINICAL TRIAL: NCT02263040
Title: A Pilot Study to Assess the Immunogenicity and Reactogenicity of High Versus Standard Dose Trivalent Inactivated Influenza Vaccine for Healthcare Workers
Brief Title: A Pilot Study to Assess the Immunogenicity and Reactogenicity of High Versus Standard Dose TIV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 14-0909
Record Dates: First submitted 2014-10-08; First posted 2014-10-13 (Estimated); Results first posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2018-08

CONDITIONS: Influenza
Keywords: influenza vaccine; adult; immunogenicity; reactogenicity
MeSH Terms: conditions — Influenza, Human | interventions — Fluzone High-Dose; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Dose Fluzone (Experimental): Fluzone High-Dose® Licensed for use in the USA in persons ≥ 65 years of age as a single dose of 0.5 mL containing 60μg hemagglutinin per virus strain
  Interventions: Biological: Fluzone High-Dose
- Fluzone (standard dose) (Active Comparator): Fluzone ® Licensed for the prevention of influenza as a single dose of 0.5 mL containing 15μg hemagglutinin per virus strain for adults
  Interventions: Biological: Fluzone (standard dose)

INTERVENTIONS:
Biological: Fluzone High-Dose — Influenza vaccine
  Arms: High Dose Fluzone
Biological: Fluzone (standard dose) — Influenza vaccine
  Arms: Fluzone (standard dose)

SUMMARY:
The objective of this pilot study is to assess the immunogenicity and reactogenicity of Fluzone High Dose with Fluzone (standard adult dose) influenza vaccines in healthcare workers.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled, observer blind trial of Fluzone High Dose trivalent inactivated influenza vaccine (HDTIV) versus Fluzone, standard dose TIV (SDTIV) in 100 healthcare workers 18-64 years of age. Participants will receive, in a 1:1 ratio, one dose of either SDTIV or HDTIV containing the strains of influenza virus as recommended by the World Health Organization for the season of recruitment. All adverse events will be collected for 7 days following the injection, serious adverse events will be collected through day 21, and serum for antibody testing will be obtained on day 0 and day 21. The primary outcome will be seroconversion to each strain of vaccine included in the vaccine, as measured by change in hemagglutination inhibition assay (HAI) titer between day 0 to day 21.

ELIGIBILITY:
Inclusion Criteria:

1. 18-64 years old, inclusive, as of October 1st of year of enrolment;
2. Healthcare worker, broadly defined as a person either providing health care, or working in an acute care hospital or long term healthcare facility;
3. Has access to email and the internet for adverse event reporting, or is willing to complete forms on paper and deliver to the site study office;
4. Understand the study, agree to its requirements, and give written consent;

Exclusion Criteria:

1. Receipt of influenza vaccine for the current northern hemisphere season prior to randomization;
2. Serious adverse event to a previous dose of influenza vaccine;
3. Immunoglobulin E mediated allergic reaction to a previous dose of influenza vaccine or to any excipients in the study vaccines
4. Previous episode of Guillain-Barré syndrome with 6 weeks of receiving an influenza vaccine;
5. Receipt of immunoglobulins, blood or blood-derived products in the past 3 months;
6. Receipt of another vaccine, or initiation of new medication, or hospital admission for any reason within the 30 days prior to the study dose of vaccine
7. Plans to receive any vaccine, initiate any medication, or be admitted to hospital before day 21 after vaccination (visit 2);
8. Known or suspected congenital or acquired immunodeficiency (including HIV infection); or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
9. Any condition, including but not limited to drug and alcohol addiction, which, in the opinion of the investigator might interfere with the ability to comply with trial conduct or completion;
10. Moderate or severe acute illness or active infection or fever (temperature ≥37.8oC) on the day the vaccine dose is due (participant may receive dose of vaccine 48 hours after symptoms have resolved and body temperature has returned to normal without the use of antipyretics.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison J McGeer, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Following publication of results

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose Fluzone: Fluzone High-Dose® Licensed for use in the USA in persons ≥ 65 years of age as a single dose of 0.5 mL containing 60μg HA per virus strain
  Fluzone High-Dose: Influenza vaccine
  Either 2014/15 OR 2015/16
- Fluzone (Standard Dose): Fluzone ® Licensed for the prevention of influenza as a single dose of 0.5 mL containing 15μg HA per virus strain for adults
  Fluzone (standard dose): Influenza vaccine
  Either: 2014/15 OR 2015/16
Period: Overall Study
Arm/Group | High Dose Fluzone | Fluzone (Standard Dose)
Started | 87 | 83
Completed | 87 | 83
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- High Dose Fluzone: Fluzone High-Dose® Licensed for use in the USA in persons ≥ 65 years of age as a single dose of 0.5mL containing 60μg HA per virus strain
  Fluzone High-Dose: Influenza vaccine
- Fluzone (Standard Dose): Fluzone ® Licensed for the prevention of influenza as a single dose of 0.5mL containing 15μg HA per virus strain for adults
  Fluzone (standard dose): Influenza vaccine
- Total: Total of all reporting groups
Arm/Group | High Dose Fluzone | Fluzone (Standard Dose) | Total
Number analyzed (Participants) | 87 | 83 | 170
Age, Continuous [Median (Full Range); unit: years] | 46 [23 to 64] | 50 [20 to 64] | 47.5 [20 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 59 | 123
  Male | 23 | 24 | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 87 | 83 | 170
Underlying chronic medical condition [Count of Participants; unit: Participants] | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Seroconversion to A/California/07/2009 (H1N1)
Description: Seroconversion to influenza strains contained in the vaccine, as measured by hemagglutination inhibition (HAI) assay. 4-fold or greater increase.
Time Frame: 21 days (18-28)
Population: A blood sample from one participant was hemolysed and not available for analysis
Measure: Count of Participants; unit: Participants
Groups:
- High Dose Fluzone: Fluzone High-Dose® Licensed for use in the USA in persons ≥ 65 years of age as a single dose of 0.5mL containing 60μg HA per virus strain
  Fluzone High-Dose: Influenza vaccine
  Either season: 2014/15 OR 2015/16
- Fluzone (Standard Dose): Fluzone ® Licensed for the prevention of influenza as a single dose of 0.5mL containing 15μg HA per virus strain for adults
  Fluzone (standard dose): Influenza vaccine
  Either season: 2014/15 OR 2015/16
Arm/Group | High Dose Fluzone | Fluzone (Standard Dose)
Number analyzed (Participants) | 86 | 83
Participants | 41 | 21

2. Primary Outcome: Number of Participants With Seroconversion to A/Texas/50/2012 (H3N2)
Description: Four-fold or higher rise in titres to A/Texas/50/2012 (H3N2) as measured by hemagglutination inhibition assay
Time Frame: 21 days post vaccination (18-28)
Measure: Count of Participants; unit: Participants
Groups:
- High Dose Fluzone: Fluzone High-Dose® Licensed for use in the USA in persons ≥ 65 years of age as a single dose of 0.5mL containing 60μg HA per virus strain
  Fluzone High-Dose: Influenza vaccine
  either 2014/15 OR 2015/16
- Fluzone (Standard Dose): Fluzone ® Licensed for the prevention of influenza as a single dose of 0.5mL containing 15μg HA per virus strain for adults
  Fluzone (standard dose): Influenza vaccine Either: 2014/15 OR 2015/16
Arm/Group | High Dose Fluzone | Fluzone (Standard Dose)
Number analyzed (Participants) | 24 | 22
Participants | 17 | 4

3. Primary Outcome: Number of Participants With Seroconversion to Influenza B/Phuket/3073/2013
Description: Four fold or higher increase in titres to B/Phuket/3073/2013 as measured by hemagglutination inhibition assay
Time Frame: 21 days post-vaccination (18-28)
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Fluzone | Fluzone (Standard Dose)
Number analyzed (Participants) | 62 | 61
Participants | 29 | 12

4. Primary Outcome: Number of Participants With Seroconversion to A/Switzerland/9715293/2013 (H3N2)
Description: Four-fold or higher rise in titres against A/Switzerland/9715293/2013 (H3N2) as measured by hemagglutination inhibition assay
Time Frame: 21 days post vaccination (18-28)
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Fluzone | Fluzone (Standard Dose)
Number analyzed (Participants) | 62 | 61
Participants | 58 | 49

5. Primary Outcome: Number of Participants With Seroconversion to B/Massachusetts/02/2012
Description: Four fold or higher increase in titres to B/Massachusetts/02/2012 as measured by hemagglutination inhibition assay
Time Frame: 21 days post-vaccination (18-28)
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Fluzone | Fluzone (Standard Dose)
Number analyzed (Participants) | 24 | 22
Participants | 8 | 3

6. Secondary Outcome: Geometric Mean Fold Ratio (GMFR) Against A/California/07/2009 (H1N1)
Description: GMFR (mean fold increase) time2/time1, as measured by hemagglutination inhibition assay
Time Frame: 21 days (18-28)
Measure: Geometric Mean (95% Confidence Interval); unit: fold ratio
Arm/Group | High Dose Fluzone | Fluzone (Standard Dose)
Number analyzed (Participants) | 86 | 83
fold ratio | 1.38 [1.28 to 1.48] | 1.20 [1.13 to 1.27]

7. Secondary Outcome: Geometric Mean Fold Ratio (GMFR): A/Switzerland/9715293/2013
Description: GMFR (mean fold increase) time2/time1, as measured by HAI titres
Time Frame: 21 days (18-28)
Measure: Geometric Mean (95% Confidence Interval); unit: fold ratio
Arm/Group | High Dose Fluzone | Fluzone (Standard Dose)
Number analyzed (Participants) | 62 | 61
fold ratio | 1.82 [1.70 to 1.94] | 1.67 [1.53 to 1.81]

8. Secondary Outcome: Geometric Mean Fold Ratio (GMFR): A/Texas/50/2012
Description: GMFR (mean fold increase) time2/time1, as measured by HAI titres
Time Frame: 21 days (18-28)
Measure: Geometric Mean (95% Confidence Interval); unit: fold ratio
Arm/Group | High Dose Fluzone | Fluzone (Standard Dose)
Number analyzed (Participants) | 24 | 22
fold ratio | 1.76 [1.36 to 2.16] | 1.15 [1.08 to 1.22]

9. Secondary Outcome: Geometric Mean Fold Ratio (GMFR): B/Phuket/3073/2013 Ether-treated
Description: GMFR (mean fold increase) time2/time1, as measured by HAI titres
Time Frame: 21 days (18-28)
Measure: Geometric Mean (95% Confidence Interval); unit: fold ratio
Arm/Group | High Dose Fluzone | Fluzone (Standard Dose)
Number analyzed (Participants) | 62 | 61
fold ratio | 1.32 [1.23 to 1.41] | 1.19 [1.11 to 1.27]

10. Secondary Outcome: Geometric Mean Fold Ratio (GMFR): B/Massachusetts/02/2012 Ether-treated
Description: GMFR (mean fold increase) time2/time1, as measured by HAI titres
Time Frame: 21 days (18-28)
Measure: Geometric Mean (95% Confidence Interval); unit: fold ratio
Arm/Group | High Dose Fluzone | Fluzone (Standard Dose)
Number analyzed (Participants) | 24 | 22
fold ratio | 1.20 [1.11 to 1.29] | 1.08 [1.02 to 1.14]

11. Secondary Outcome: Number of Participants Reporting Adverse Event: Injection Site
Description: Any local adverse event following immunization,self reported in daily diary Includes the maximum values for any one of: redness, warmth, swelling, or bruising
Time Frame: 7 days
Population: All participants were able to provide data
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Fluzone | Fluzone (Standard Dose)
Number analyzed (Participants) | 87 | 83
Participants
  none | 47 | 62
  mild | 34 | 21
  moderate | 6 | 0

12. Secondary Outcome: Number of Participants Reporting Adverse Event: Systemic
Description: Any systemic adverse event following immunization,self reported in daily diary Includes the maximum value reported for any one of: myalgia, arthralgia, headache, malaise, fatigue, weakness, sweating, shivering, or feverishness
  Defined as:
  None: Not at all Mild: Present, but did not interfere with activities Moderate: Interfered with activities, but didn't prevent them Extreme: Prevented activities
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Fluzone | Fluzone (Standard Dose)
Number analyzed (Participants) | 87 | 83
Participants
  None | 41 | 42
  Mild | 23 | 25
  Moderate | 18 | 13
  Extreme | 5 | 3

ADVERSE EVENTS:
Time Frame: 6 months
Description: Daily diary for 7 days Nursing note at day 21 Asked to report to clinic for 6 months after vaccination
Arm/Group | High Dose Fluzone | Fluzone (Standard Dose)
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/83
Other Adverse Events (participants affected / at risk) | 26/87 | 6/83
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Fluzone (N=87) | Fluzone (Standard Dose) (N=83)
Myalgia (General disorders) | 13 (13) | 6 (6) — Moderate or extreme: interfered with, or prevented, daily activities
Headache (General disorders) | 8 (8) | 4 (4) — Moderate or extreme: interfered with, or prevented, daily activities
Fatigue (General disorders) | 9 (9) | 6 (6) — Moderate or extreme: interfered with, or prevented, daily activities
Malaise (General disorders) | 5 (5) | 4 (4) — Moderate or extreme: interfered with, or prevented, daily activities

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No